CLINICAL TRIAL: NCT01959945
Title: Evaluation of the Safety, Reactogenicity and Immunogenicity of Flublok Quadrivalent (Quadrivalent Recombinant Influenza Vaccine,Seasonal Formulation) Administered Intramuscularly to Healthy Children and Adolescents Age 6-17 Years
Brief Title: Safety, Reactogenicity and Immunogenicity of Flublok Quadrivalent (Recombinant Influenza Vaccine,Seasonal Formulation)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PSC08
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study Group 1, Flublok (Experimental): Participants at 9 years to 17 years of age at enrollment, Flublok® Quadrivalent Influenza Virus Vaccine
  Interventions: Biological: Flublok® Quadrivalent Influenza Virus Vaccine
- Study Group 2, Fluarix (Active Comparator): Participants at 9 years to 17 years of age at enrollment, Fluarix Quadrivalent® Influenza Virus Vaccine
  Interventions: Biological: Fluarix Quadrivalent® Influenza Virus Vaccine
- Study Group 3, Flublok (Experimental): Participants at 6 years to 8 years of age at enrollment, Flublok® Quadrivalent Influenza Virus Vaccine
  Interventions: Biological: Flublok® Quadrivalent Influenza Virus Vaccine
- Study Group 4, Fluarix (Active Comparator): Participants at 6 years to 8 years of age at enrollment, Fluarix Quadrivalent® Influenza Virus Vaccine
  Interventions: Biological: Fluarix Quadrivalent® Influenza Virus Vaccine

INTERVENTIONS:
Biological: Flublok® Quadrivalent Influenza Virus Vaccine — Intramuscular (Relevant year formulation)
  Other Names: Recombinant Influenza Vaccine (RIV4); Flublok Influenza Vaccine; rHA; rHA0; Recombinant Hemagglutinin
  Arms: Study Group 1, Flublok; Study Group 3, Flublok
Biological: Fluarix Quadrivalent® Influenza Virus Vaccine — Intramuscular (Relevant year formulation)
  Arms: Study Group 2, Fluarix; Study Group 4, Fluarix

SUMMARY:
Flublok was studied previously in children 6 -59 months of age and demonstrated less than satisfactory immunogenicity results, especially in the 6-36 month age group. Thus, the initial introduction of Flublok Quadrivalent Formulation (RIV4) into the pediatric population will evaluate immunogenicity and safety older children and adolescents, aged 6-17. This clinical trial is designed to demonstrate safety and non-inferior immunogenicity of Flublok-Q in pediatric subjects 6-17 years of age as compared to IIV4. Positive results in this study may support further studies in younger children.

DETAILED DESCRIPTION:
The U.S. Advisory Committee on Immunization Practices (ACIP) recommends that all people ≥6 months of age receive influenza vaccine annually. Recommendations for influenza immunization of children vary somewhat among countries in the European Union, but immunization of children at high risk for complications of influenza infection is recommended by WHO and according to criteria in most countries. Currently, the immunization practices are progressing to quadrivalent formulations of inactivated influenza vaccines (IIV4) which are approved in the US for most of the indicated population. Additionally, live attenuated vaccine (LAIV4) is approved in the U.S. for individuals aged 2-49 years and Flublok®(RIV3), a purified trivalent recombinant hemagglutinin protein vaccine is approved in the U.S. for adults 18-49 years of age. Children are at particular risk of complications of influenza, including the B lineages, so expansion of the Flublok indication into the pediatric age group with a quadrivalent formulation is warranted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 6-17 years (Cohort A: 6-8 years of age; Cohort B: 9-17 years of age)
2. Female subjects of child-bearing potential (as defined by the onset of menses) must agree to avoid becoming pregnant and to use effective method of contraception or practice abstinence for at least 28 day prior to the first study vaccine administration, until the completion of the study. Female subjects of child-bearing potential must have a negative pregnancy test within 24 hours prior to vaccine administration.
3. In good general health, as determined by medical history and targeted physical examination, if indicated

The parent(s) or legal representative(s) of each potential subject must:

1. Comprehend the study requirements and agree to comply with planned study procedures and visits
2. Provide written consent prior to enrollment and initiation of any study procedures Pediatric assent will be obtained in accordance with the Institutional Review Board/Independent Ethics Committee determination.

Exclusion Criteria:

1. Known allergy to eggs, severe allergy (e.g. anaphylaxis) to other components of either vaccine or contraindications to receipt of the comparator IIV4
2. Immunosuppression as a result of an underlying illness or treatment. Note: Subjects on nasal or topical steroids will be allowed
3. Active neoplastic disease or a history of any malignancy.
4. History of receiving influenza vaccine within the past 6 months or plans during the study to receive influenza vaccine outside of this study.
5. History of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
6. Receipt of any non-study licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study, or plans during the study to receive a licensed vaccine within 4 weeks of a study dose [See above for influenza vaccines].
7. Acute or chronic medical condition that, in the opinion of the investigator, would render immunization unsafe or would interfere with the evaluation of immune responses
8. History of severe reactions following immunization.
9. An acute illness, including a body temperature greater than 100*F, within 3 days prior to immunization.
10. Receipt of an experimental vaccine or medication within 1 month prior to enrollment in this study, or expectation of receiving an experimental vaccine, medication, or blood product during the study Stage in which the subject will participate.
11. Developmental delay, neurologic disorder, or seizure disorder requiring ongoing medical management (note: history of seizure is not an exclusion criterion).
12. Any other condition or situation that would, in the opinion of the investigator, place the potential subject an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
13. History of Guillain-Barré syndrome.
14. Known pregnancy, positive urine or serum pregnancy test within 24 hours prior to planned study vaccination, or breast-feeding.
15. Concurrent participation in another clinical trial (in active or follow-up phase).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 219 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Dunkle, MD, Study Chair — Protein Sciences Corporation
Locations (1):
- Maine Research Associates, LLC, Auburn, Maine, United States

REFERENCES:
- [Derived] Dunkle LM, Izikson R, Patriarca PA, Goldenthal KL, Cox M, Treanor JJ. Safety and Immunogenicity of a Recombinant Influenza Vaccine: A Randomized Trial. Pediatrics. 2018 May;141(5):e20173021. doi: 10.1542/peds.2017-3021. Epub 2018 Apr 2. PMID 29610401
- See also: Related Info — http://www.proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The randomized population (219 subjects) includes all subjects who were randomized and the safety population (217 subjects) includes all randomized subjects who received any dose of study vaccine and provided any safety. Two (2) randomized subjects did not fit the criteria to be included in the safety population and were excluded from the analysis.
Groups:
- Study Group 1, Flublok Cohort A: Participants at 9 years to 17 years of age at enrollment, Flublok® Quadrivalent Influenza Virus Vaccine
  Flublok® Quadrivalent Influenza Virus Vaccine: Intramuscular (Relevant year formulation)
- Study Group 2, Fluarix Cohort A: Participants at 9 years to 17 years of age at enrollment, Fluarix Quadrivalent® Influenza Virus Vaccine
  Fluarix Quadrivalent® Influenza Virus Vaccine: Intramuscular (Relevant year formulation)
- Study Group 3, Flublok Cohort B: Participants at 6 years to 8 years of age at enrollment, Flublok® Quadrivalent Influenza Virus Vaccine
  Flublok® Quadrivalent Influenza Virus Vaccine: Intramuscular (Relevant year formulation)
- Study Group 4, Fluarix Cohort B: Participants at 6 years to 8 years of age at enrollment, Fluarix Quadrivalent® Influenza Virus Vaccine
  Fluarix Quadrivalent® Influenza Virus Vaccine: Intramuscular (Relevant year formulation)
Period: Overall Study
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 2, Fluarix Cohort A | Study Group 3, Flublok Cohort B | Study Group 4, Fluarix Cohort B
Started | 80 | 78 | 28 | 31
Completed | 76 | 75 | 9 | 15
Not Completed | 4 | 3 | 19 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 2, Fluarix Cohort A | Study Group 3, Flublok Cohort B | Study Group 4, Fluarix Cohort B | Total
Number analyzed (Participants) | 80 | 78 | 28 | 31 | 217
Age, Customized [Number; unit: participants]
  9-17 years | 80 | 78 | 0 | 0 | 158
  6-8 years | 0 | 0 | 28 | 31 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 17 | 12 | 111
  Male | 38 | 38 | 11 | 19 | 106
Region of Enrollment [Number; unit: participants]
  United States | 80 | 78 | 28 | 31 | 217

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Events and Unsolicited Adverse Events Following Vaccination With Quadrivalent Vaccine.
Description: Solicited injection site reactions: Pain, Bruising, Redness, and Swelling; Solicited systemic reactions: Headache, Chills, Fever, Fatigue, Muscle Pain, Joint Pain and Nausea.
Time Frame: Day 0 up to Day 28 post vaccination
Measure: Number; unit: participants
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 3, Flublok Cohort B | Study Group 2, Fluarix Cohort A | Study Group 4, Fluarix Cohort B
Number analyzed (Participants) | 80 | 28 | 78 | 31
participants
  Solicited Systemic Events | 47 | 16 | 53 | 18
  Solicited Local Events | 39 | 14 | 42 | 14
  Unsolicited Adverse Events | 19 | 13 | 26 | 15

2. Secondary Outcome: Geometric Mean Titers of Antibodies to Vaccine Antigens Following Vaccination With Quadrivalent Vaccine
Description: Immunogenicity will be evaluated prior to vaccination and at 28 days after vaccination using the hemagglutination inhibition (HAI) technique. For each influenza vaccine strain, pre and post vaccination geometric mean titers (GMTs) and seroprotection and seroconversion will be calculated.
Time Frame: Day 0 and Day 28 after final vaccination (Cohort B includes 1-Dose subjects at Day 28 and 2-Dose subjects at Day 56)
Population: The evaluable immunogenicity population includes randomized subjects who received the assigned number of doses of study vaccine and have HAI titers available from blood draws taken at baseline and ~28 days following completion of immunization (~Day 56 for 2-dose subjects), which accounts for the discrepancy in Participants Analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 2, Fluarix Cohort A | Study Group 3, Flublok Cohort B | Study Group 4, Fluarix Cohort B
Number analyzed (Participants) | 75 | 77 | 26 | 28
titer
  Day 0 - A/California/7/2009 | 54.94 [38.83 to 77.73] | 59.79 [43.05 to 83.02] | 85.89 [44.83 to 164.57] | 57.04 [31.29 to 103.98]
  Day 28 - A/California/7/2009 | 914.92 [693.4 to 1207.19] | 564.23 [449.6 to 708.07] | 1224.31 [749.8 to 1999.05] | 695.03 [501.5 to 963.32]
  Day 0 - A/Texas/50/2012 | 181.57 [140.4 to 234.83] | 141.91 [108.7 to 185.25] | 272.74 [181.7 to 409.37] | 161.32 [113.0 to 230.37]
  Day 28 - A/Texas/50/2012 | 852.30 [698.1 to 1040.64] | 531.36 [449.8 to 627.75] | 1071.58 [776.2 to 1479.45] | 629.48 [451.4 to 877.78]
  Day 0 - B/Massachusetts/2/2012 | 20.44 [16.11 to 25.94] | 21.17 [16.15 to 27.75] | 13.89 [9.54 to 20.23] | 12.19 [8.89 to 16.72]
  Day 28 - B/Massachusetts/2/2012 | 161.02 [124.8 to 207.83] | 119.96 [95.07 to 151.37] | 111.14 [69.87 to 176.79] | 122.90 [81.92 to 184.38]
  Day 0 - B/Brisbane/60/2008 | 12.49 [10.17 to 15.33] | 10.56 [8.62 to 12.94] | 11.43 [8.32 to 15.69] | 9.36 [7.05 to 12.43]
  Day 28 - B/Brisbane/60/2008 | 51.73 [39.73 to 67.34] | 59.67 [47.30 to 75.27] | 73.82 [45.05 to 120.96] | 60.74 [40.35 to 91.42]

3. Secondary Outcome: Seroconversion to Vaccine Antigens Following Vaccination With Quadrivalent Vaccine
Description: Seroconversion is defined as: Either a pre vaccination titer < 10 (1/dil) and a post vaccination titer ≥ 40 (1/dil), or a pre vaccination titer ≥ 10 (1/dil) and a ≥ 4 fold increase in post vaccination titer at Day 28 after the final vaccination.
Time Frame: Day 28 after final vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 2, Fluarix Cohort A | Study Group 3, Flublok Cohort B | Study Group 4, Fluarix Cohort B
Number analyzed (Participants) | 75 | 77 | 26 | 28
percentage of participants
  H1N1: A/California/07/2009 | 87 [76.8 to 93.4] | 68 [55.9 to 77.8] | 88 [69.8 to 97.6] | 75 [55.1 to 89.3]
  H3N2: A/Texas/50/2012 | 59 [46.7 to 69.9] | 49 [37.8 to 61.0] | 54 [33.4 to 73.4] | 50 [30.6 to 69.4]
  B/Massachusetts/2/2012 | 69 [57.6 to 79.5] | 61 [49.2 to 72.0] | 77 [56.4 to 91.0] | 82 [63.1 to 93.9]
  B/Brisbane/60/2008 | 52 [39.4 to 65.1] | 67 [53.7 to 78.0] | 69 [48.2 to 85.7] | 73 [52.2 to 88.4]

4. Secondary Outcome: Seroprotection to Vaccine Antigens Following Vaccination With Quadrivalent Vaccine
Description: Seroprotection is defined as: A titer ≥ 40 (l/dil) at pre vaccination and at Day 28 after the final vaccination.
Time Frame: Day 28 after final vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 2, Fluarix Cohort A | Study Group 3, Flublok Cohort B | Study Group 4, Fluarix Cohort B
Number analyzed (Participants) | 75 | 77 | 26 | 28
percentage of participants
  H1N1: A/California/07/2009 | 97 [90.7 to 99.7] | 99 [93.0 to 100.0] | 100 [86.8 to 100.0] | 100 [87.7 to 100.0]
  H3N2: A/Texas/50/2012 | 100 [95.2 to 100.0] | 100 [95.3 to 100.0] | 100 [86.8 to 100.0] | 100 [87.7 to 100.0]
  B/Massachusetts/2/2012 | 91 [81.7 to 96.2] | 90 [80.6 to 95.4] | 85 [65.1 to 95.6] | 89 [71.8 to 97.7]
  B/Brisbane/60/2008 | 78 [65.5 to 87.3] | 86 [74.6 to 93.3] | 85 [65.1 to 95.6] | 81 [60.6 to 93.4]

ADVERSE EVENTS:
Time Frame: All AEs collected 28 days after final study immunization and all Serious Adverse Events (SAEs) collected through one (1) year after last study immunization.
Arm/Group | Study Group 1, Flublok Cohort A | Study Group 3, Flublok Cohort B | Study Group 2, Fluarix Cohort A | Study Group 4, Fluarix Cohort B
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/28 | 0/78 | 1/31
Other Adverse Events (participants affected / at risk) | 9/80 | 10/28 | 14/78 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group 1, Flublok Cohort A (N=80) | Study Group 3, Flublok Cohort B (N=28) | Study Group 2, Fluarix Cohort A (N=78) | Study Group 4, Fluarix Cohort B (N=31)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — A 9 year old African American male with a medical history of asthma was hospitalized for one day for treatment of an asthma attack that occurred 5 months after receipt of IIV4 study vaccine. The event was considered not related to study vaccine.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study Group 1, Flublok Cohort A (N=80) | Study Group 3, Flublok Cohort B (N=28) | Study Group 2, Fluarix Cohort A (N=78) | Study Group 4, Fluarix Cohort B (N=31)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Injection site erythema (General disorders) | 2 | 1 | 0 | 1
Injection site pain (General disorders) | 1 | 2 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 4
Viral infection (Infections and infestations) | 1 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 4 | 0

LIMITATIONS AND CAVEATS:
The numbers of subjects available for analysis in Cohort B (age 6-8 years) was fewer than anticipated due to early termination of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less